CLINICAL TRIAL: NCT04259801
Title: Investigation of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of NNC0480-0389 in Combination With Semaglutide s.c.
Brief Title: First Research Study to Look at How Two Medicines, NNC0480-0389 and Semaglutide, Work Together in Healthy People, in People With High Body Weight and in People With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9389-4536; 2019-002857-44 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1236-4114 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers; Overweight; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Part 1: Single ascending dose Part 2: Multiple ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NNC0480-0389 and semaglutide (Experimental): Part 1: 6 subjects will receive a single subcutaneous (s.c., under the skin) dose of NNC0480-0389 co-administered with s.c. semaglutide.
  Part 2: 12 subjects will receive 4 doses of s.c. NNC0480-0389 co-administered with s.c. semaglutide, after 8 weeks of dosing with s.c semaglutide.
  Interventions: Drug: NNC0480-0389; Drug: Semaglutide
- NNC0480-0389 and placebo (semaglutide) (Experimental): Part 1: 4 subjects will receive a single dose of s.c. NNC0480-0389 co-administered with semaglutide placebo.
  Part 2: 4 subjects will receive 4 doses of s.c. NNC0480-0389, co-administered with semaglutide placebo after 8 weeks of dosing with semaglutide placebo.
  Interventions: Drug: NNC0480-0389; Drug: Placebo (NNC0480-0389)
- Placebo (NNC0480-0389) with semaglutide (Active Comparator): Part 1: 2 subjects will receive a single dose of placebo (NNC0480-0389), co-administered with s.c. semaglutide.
  Part 2: 4 subjects will receive 4 doses of placebo (NNC0480-0389), co-administered with s.c. semaglutide, after 8 weeks of dosing with s.c. semaglutide
  Interventions: Drug: Semaglutide; Drug: Placebo (semaglutide)
- Placebo (NNC0480-0389) with placebo (semaglutide) (Placebo Comparator): Part 1: 3 subjects will receive a single dose of placebo (NNC0480-0389), co-administered with semaglutide placebo.
  Part 2: 2 subjects will receive 4 doses of placebo (NNC0480-0389), co-administered with semaglutide placebo, after 8 weeks of dosing with semaglutide placebo.
  Interventions: Drug: Placebo (NNC0480-0389); Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: NNC0480-0389 — Part 1: A single dose of NNC0480-0389, dose increased in each cohort. Part 2: Weekly doses (for 4 weeks) of NNC0480-0389, dose increased in each cohort.
  Arms: NNC0480-0389 and placebo (semaglutide); NNC0480-0389 and semaglutide
Drug: Semaglutide — Part 1: Single dose of semaglutide (0.5 mg). Part 2: Weekly doses of semaglutide alone for 8 weeks (2 x 0.25 mg, 2 x 0.5 mg and 4 x 1 mg) followed by weekly fixed doses of 1 mg semaglutide for 4 weeks.
  Arms: NNC0480-0389 and semaglutide; Placebo (NNC0480-0389) with semaglutide
Drug: Placebo (NNC0480-0389) — Placebo for NNC0480-0389. Part 1: A single dose of placebo (NNC0480-0389), dose increased in each cohort. Part 2: Weekly doses (for 4 weeks) of placebo A, dose increased in each cohort.
  Arms: NNC0480-0389 and placebo (semaglutide); Placebo (NNC0480-0389) with placebo (semaglutide)
Drug: Placebo (semaglutide) — Part 1: Single dose of placebo (semaglutide) (0.5 mg). Part 2: Weekly doses of placebo (semaglutide) alone for 8 weeks (2 x 0.25 mg, 2 x 0.5 mg and 4 x 1 mg) followed by weekly fixed doses of 1 mg semaglutide for 4 weeks.
  Arms: Placebo (NNC0480-0389) with placebo (semaglutide); Placebo (NNC0480-0389) with semaglutide

SUMMARY:
The purpose of this study is to investigate how safe, and how well tolerated, the new study drug NNC0480-0389 is when it is given together with semaglutide. This will be investigated in healthy participants, participants with high bodyweight and participants with type 2 diabetes (T2D). NNC0480-0389 has not been given to humans before. It has been previously tested in the laboratory and on animals. NNC0480-0389 will be tested at various dose levels. Semaglutide is a new approved drug and is already available on the market for treatment of diabetes. It will also be investigated how quickly and to what extent NNC0480-0389 and semaglutide are taken up and eliminated from the body. This is called pharmacokinetics. The effect of NNC0480-0389 given together with semaglutide will also be investigated on body weight and glucose levels in the blood. This is called pharmacodynamics. The effects of NNC0480-0389 and/or semaglutide will be compared to the effects of a placebo. A placebo is a "dummy" medicine without any active medicine. Placebo looks like NNC0480-0389 and/or semaglutide. There are 4 possibilities for which treatment participants will get; participants will receive NNC0480-0389 and semaglutide or NNC0480-0389 and placebo or placebo with semaglutide, or placebo with placebo. Participants and the responsible doctor will not know which combination participants will be given. This is called a double-blinded study. However, this information can be looked up during the study if it is important for participants' health. The study medicines will be given as injections under the skin. Participants will be in the study for about 25 weeks.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Male aged 18-45 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 kg/m^2 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Part 2 (not applicable for proof-of-concept (PoC) cohort):

* Body mass index between 20.0 kg/m^2 and 39.9 kg/m^2 (both inclusive).
* Female of non-childbearing potential or male aged 18-55 years (both inclusive) at the time of signing informed consent.
* Considered to be eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Part 2 (only applicable for PoC cohort):

* Body mass index between 25.0 kg/m^2 and 39.9 kg/m^2 (both inclusive). Overweight or obesity should be due to excess adipose tissue, as judged by the investigator.
* Female of non-childbearing potential or male aged 18-64 years (both inclusive) at the time of signing informed consent.
* Considered to be eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Diagnosed with type 2 diabetes at least 90 days prior to the day of screening.
* Subjects treated with diet and exercise as monotherapy or in combination with 1-2 of the following anti-diabetic drug(s) at a stable dose for at least 30 days prior to screening: metformin, sulfonylureas, meglitinides, DPP-4 inhibitors, alpha-glucosidase inhibitors, thiazolidinediones, GLP-1 receptor agonists or SLGT-2 inhibitors. The metformin dose should be between 1500 mg to 3000 mg or maximum tolerated or effective dose documented in subject's medical record.
* Glycosylated haemoglobin (HbA1c) in the range of 6.5% (inclusive) and 10% (non-inclusive).

Exclusion Criteria:

Part 1:

* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* HbA1c equal to or above 6.5 % (48 mmol/mol) at screening.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, occasional use of acetaminophen, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation within 14 days prior to the day of screening. Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.

Part 2 (not applicable for PoC cohort):

* Any disorder (except for conditions associated with T2D for the PoC cohort) which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions (except conditions associated with T2D for PoC Cohort).
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, occasional use of acetaminophen, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation within 14 days prior to the day of screening.
* HbA1c equal to or above 6.5 % (48 mmol/mol) at screening.

Part 2 (only applicable for PoC cohort):

* Any disorder (except for conditions associated with T2D for the PoC cohort) which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, or endocrinological conditions (except conditions associated with T2D for PoC Cohort).
* Use of any prohibited medications as listed in the protocol within 14 days of screening.
* Use of prescribed medications at the time of screening at a dose that had not been stable within 30 days prior to screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) in Part 1 | From time of dosing (day 1) until completion of follow-up visit (day 71)
  Number of events
Number of treatment emergent adverse events (TEAE) in Part 2 | From first combination dosing (day 57) until completion of follow-up visit (day 148)
  Number of events

SECONDARY OUTCOMES:
Area under the NNC0480-0389 plasma concentration-time curve from time | From baseline (day 1) to post treatment follow-up (day 71)
  h∙nmol/L
Maximum plasma concentration of NNC0480-0389 after administration of a single dose | From baseline (day 1) to post treatment follow-up (day 71)
  nmol/L
Area under the semaglutide plasma concentration time curve from time of dosing to infinity after administration of a single dose | From baseline (day 1) to post treatment follow-up (day 71)
  h∙nmol/L
The maximum concentration of semaglutide after administration of a single dose | From baseline (day 1) to post treatment follow-up (day 71)
  nmol/L
Area under the NNC0480-0389 plasma concentration-time curve from 0 to 168 hours after administration of the 4th dose of NNC0480-0389 in week 12 | From administration of dose in week 12 (day 78) to day 85
  h∙nmol/L
Maximum plasma concentration of NNC0480-0389 after administration of the 4th dose of NNC0480-0389 in week 12 | From administration of dose in week 12 (day 78) to post treatment follow-up (day 148)
  nmol/L
Area under the semaglutide plasma concentration-time curve from 0-168 hours after administration of the 12th dose of semaglutide | From administration of dose in week 12 (day 78) to day 85
  h∙nmol/L
The maximum concentration of semaglutide after administration of the 12th dose of semaglutide | From administration of dose in week 12 (day 78) to post treatment follow-up (day 148)
  nmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com